CLINICAL TRIAL: NCT03858114
Title: Active Ageing and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Mauro Giovanni Carta, Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PG/2018/15546
Record Dates: First submitted 2019-02-13; First posted 2019-02-28 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Aging; Chronic Disease; Cognitive Decline; Quality of Life; Physical Activity
MeSH Terms: conditions — Chronic Disease; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild-to-moderate physical activity (Experimental): Three sessions/week, for 12 weeks, of mild-to-moderate physical activity, of mixed type (aerobic-anaerobic), supervised by expert and qualified personnel (physical education instructors) and performed in a gym.
  Interventions: Other: Mild-to-moderate physical activity
- Cultural group program (Active Comparator): Cultural group program with thematic meetings and one visit/week to places of historical and artistic interest in the city of Cagliari, Sardinia, accompanied by expert guides (accredited tour guides).
  Interventions: Other: Cultural group program

INTERVENTIONS:
Other: Mild-to-moderate physical activity — According to ACSM guidelines, mild-to-moderate Physical Activity (PA) will be established as ≤ 60% of the Heart Rate Reserve (HRR). Baseline HR will be registered for all participants for three days, and the mean data will be utilized. PA intervention will consist of three phases:
  1. warm up (10 minutes), up to 40% of HRR, with slow, dynamic movements and stretching for principal muscular groups;
  2. Active phase (45 minutes), from >40% to 60% HRR, with static and dynamic exercises for postural control and spine mobility, and balance exercises, with activation of core muscles;
  3. cool down (10 minutes), < 40% of HRR, with cardiorespiratory cool-down exercises followed by relaxation, and post-stretch exercises to return muscles to a pre-exercises length.
  Arms: Mild-to-moderate physical activity
Other: Cultural group program — A cultural group program with 12-weeks thematic meetings on places of historical and artistic interest in the city of Cagliari, Sardinia, with one visit/week to the same sites. The participants will be accompanied by expert tour guides to museums, monuments, city parks and archeological sites.
  Arms: Cultural group program

SUMMARY:
Background: 36% of the Italian population will have more than 65 years in 2050. The European Union has indicated among its priorities to increase research on active aging. Physical activity contrasts disability linked to chronic diseases, has positive effects on the quality of life and on biological rhythms, prevents the decline of motor functions, improves the immune response, and prevents / positively affects metabolic disorders. It also provides valuable support in coping with cognitive decline and memory, and acts on depressive symptomatology.

The literature on active aging is based, to date, on studies with small samples, rarely conducted with a randomized controlled method, whose outcomes often appear contradictory.

The multidisciplinary project the investigators propose is an opportunity to address the issues mentioned above and to acquire further knowledge in the field of active aging.

Objectives: the main objective of the study is to evaluate the effects of mild-to-moderate physical activity in a sample of over-65 years-old persons, on Quality of Life, and on biomechanical parameters (static-dynamic balance, mobility). The secondary objectives are aimed at assessing whether a protocol of mild-to-moderate physical activity can improve:

* Metabolic functions
* Cognitive performance
* Perception of pain
* Social rhythms and psychological wellbeing
* Inflammatory state Design: randomized controlled trial (RCT), single-blinded, with follow-up.

Sample: participants will be ≥ 65 years old, of both genders, sedentary, enrolled in two arms through a random assignment (treatment/control) with ratio of 1:1, as following:

* about 60 subjects who will carry out a light-to-moderate physical activity intervention (experimental group);
* about 60 subjects in the control group, who will participate in group cultural activities (active comparison group).

Assessment: the assessment will include socio-demographic variables; variables of psychophysical wellbeing; cognitive variables; variables related to physical health; biomechanical variables; assessment of skin integrity; lab tests on blood samples.

Times of evaluations: both groups will be subjected to the measurements of the present study according to the following schedule:

* T0 (baseline): before the start of the intervention
* T1: 12 weeks after T0 (at the end of the intervention)
* T2: after 20 weeks from T0 (follow up 1)
* T3: 48 weeks after T0 (follow-up 2).

ELIGIBILITY:
Inclusion Criteria:

* sedentary (do not practicing regular physical activity, at least 2 times a week, for at least 6 months).
* certificate of fitness for non-competitive physical activity issued by a specialist in Sports Medicine.

Exclusion Criteria:

* BMI (Body Mass Index)>35;
* severe cardiovascular disease, such as myocardial infarction in the previous 2 years, aorto-coronary bypass, pacemaker or mechanical valvular prosthesis, aortic stenosis, acute pericarditis, acute myocarditis, aneurysms, angina, arrhythmias, moderate or severe aortic and mitral valve failure, arterial pressure at rest: systolic> 200 mmHg, or diastolic> 100 mmHg, pharmacologically non-compensated chronic atrial fibrillation, treatment with oral anticoagulants, thrombophlebitis or pulmonary embolism in the previous 2 years, ongoing moderate/severe anemia (Hb <10 mg / dL);
* serious problems of autonomous walking, such as fractures of the lower limbs in the previous 2 years, upper limb fractures in the previous 6 months, surgical interventions (non-arthroscopic) in the joints in the previous 2 years, any reason of absolute immobility for more than a week in the previous two months, and for more than two weeks in the previous 6 months, severe osteoporosis, walking problems (eg, use of crutches or stick);
* severe metabolic disorders, such as insulin-treated diabetes mellitus or with HbA1c > 8, or pharmacologically non-compensated thyreopathies (hyper/hypothyroidism);
* severe neurological conditions that determine the impossibility to carry out the physical activity protocol, such as stroke cerebri in the previous 2 years, or Parkinson's disease;
* severe bronchopulmonary disorders, such as severe bronchial asthma, severe chronic obstructive pulmonary disease, or pulmonary emphysema;
* severe renal disorders and make dialysis;
* severe glaucoma or retinal detachment in the previous 3 months;
* malignant neoplasm in progress, or in the previous 2 years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-11-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline Short Form Health Survey 12-items (SF-12) score at 12 weeks. | Baseline (T0), and change from baseline at twelve (T1) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on Quality of Life, measured by the Short Form Health Survey 12-items (SF-12). SF-12 measures perceived Quality of Life, with higher scores corresponding to a better subjective perception of Quality of Life, and can be aggregated as Physical Component score (ranging from 6 to 18), Mental Component score (ranging from 6 to 25), and summed as Global Component score (ranging from 12 to 43).
Change from baseline Short Form Health Survey 12-items (SF-12) score at 20 weeks. | Baseline (T0), and change from baseline at twenty (T2) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on Quality of Life, measured by the Short Form Health Survey 12-items (SF-12). SF-12 measures perceived Quality of Life, with higher scores corresponding to a better subjective perception of Quality of Life, and can be aggregated as Physical Component score (ranging from 6 to 18), Mental Component score (ranging from 6 to 25), and summed as Global Component score (ranging from 12 to 43).
Change from baseline Short Form Health Survey 12-items (SF-12) score at 48 weeks. | Baseline (T0), and change from baseline at forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on Quality of Life, measured by the Short Form Health Survey 12-items (SF-12). SF-12 measures perceived Quality of Life, with higher scores corresponding to a better subjective perception of Quality of Life, and can be aggregated as Physical Component score (ranging from 6 to 18), Mental Component score (ranging from 6 to 25), and summed as Global Component score (ranging from 12 to 43).
Change in gait speed measured using inertial sensor | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on mobility, assessed by changes in gait speed measured using a single wearable inertial sensor located in the low back (L4-L5 vertebrae)
Change in functional balance measured using inertial sensor | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on functional balance, assessed by changes in time needed to complete a 3m Timed-up-and-go (TUG) test. This will be carried out using a single wearable inertial sensor located in the low back (L4-L5 vertebrae)

SECONDARY OUTCOMES:
Change in anthropometric measurements: BMI | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on BMI (Body Mass Index), measured as the body weight divided by the square of the body height (kg/ m2).
Change in anthropometric measurements: waist circumference | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on waist circumference, measured in centimeters.
Change in body composition | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on body composition (e.g. lean and fat mass, and total body water), measured by bioimpedentiometry.
Change in cognitive status. | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on cognitive functions, assessed by the Addenbrooke's Cognitive Examination Revised (ACE-R), which contains 5 sub-scores, each one representing one cognitive domain: attention/orientation (18 points), memory (26 points), fluency (14 points), language (26 points) and visuospatial (16 points). ACE-R maximum score is 100, composed by the addition of the all domains.
Change in inflammatory status: blood cells count. | Baseline (T0), and change from baseline at twelve (T1) and twenty (T2) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on inflammatory status, measured by lab analyses (CBC + fl. + Plt), measured by blood cells count (e.g. erythrocytes count, total and differential leucocytes count, platelets count), measured as number of cells/microliter. The normal red blood cells (RBC) range for men is 4.7 to 6.1 million cells/mcL, for women is 4.2 to 5.4 million mcL. The normal white blood cells (WBCs) count ranges 5000-10000/mcL, with normal percentages of WBCs types as following: 55-73% neutrophils, 20-40% lymphocytes, 2-8% monocytes, 1-4% eosinophils, 0.5-1% basophils. The normal platelets count ranges 150000-450000/mcL.
Change in inflammatory status: erythrocyte sedimentation rate. | Baseline (T0), and change from baseline at twelve (T1) and twenty (T2) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on inflammatory status, measured by erythrocyte sedimentation rate (ESR). The normal range is 0-22 millimeters/hour for men and 0-29 millimeters/hour for women.
Change in inflammatory status: C-reactive proteine. | Baseline (T0), and change from baseline at twelve (T1) and twenty (T2) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on inflammatory status, measured by C-reactive proteine (CRP). Normal concentrations of CRP varies between 0.8 mg/L to 3.0 mg/L.
Change in metabolic status: basal glycaemia. | Baseline (T0), and change from baseline at twelve (T1) and twenty (T2) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on metabolic status, measured by basal glycaemia, ranging from 72 to 99 mg/dL.
Change in metabolic status: blood lipids. | Baseline (T0), and change from baseline at twelve (T1) and twenty (T2) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on metabolic status, measured as blood lipids concentration (mg/dL) for Total cholesterol (limit value: 199 mg/dL) , HDL cholesterol (normal value men: 41-59 mg/dL; normal value women: 51-60 mg/dL), Triglycerides (normal value: 150-199 mg/dL).
Change in psychological wellbeing | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on depressive/anxiety symptoms, assessed by the Patient Health Questionnaire-9 items (PHQ-9) questionnaire. The PHQ-9 ranges from 0 (no psychopathological symptoms, better score) to 27 (worse score), with minor depression cut-off for scores ≥5, and major depressive disorder cut-off scores ≥10.
Change in social rhythms | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on social rhythms, assessed by the Brief Social Rhythms Scale (BSRS) questionnaire. The BSRS consists of ten items, assessing the general regularity with which interviewed engage in basic daily activities during the workweek and on the weekend, ranging from 1 (very regularly) to 6 (very irregularly), with high mean scores indicating high irregularity. Summary scores are the average across all 10 items.
Change in disability perception | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on physical disability perception, measured by the Sickness Impact Profile-Roland (SIP-Roland) scale for disability. The SIP-Roland scale is a 23-items questionnaire with a total score ranging from 0 (better score, no disability) to 23 (worse score).
Change in pain perception | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on physical pain perception, measured by the NPRS (Numeric Pain Rating Scale). The NPRS is a visual-analogic scale rating the current pain perception, ranging from 0 (better score, no pain) to 10 (the worst pain imaginable).
Change in wrinkles severity | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on wrinkles severity, measured by Visual Wrinkles Scale, assessing the wrinkles grade ranging from 0 (no wrinkles) to 5 (very deep wrinkle, redundant fold) in the following anatomic points: horizontal forehead lines, glabellar frown lines, periorbital lines, preauricular lines, cheek lines, naso-labial folds, radial upper and lower lip lines, corner of the mouth lines, "marionette lines", labiomental crease, horizontal neck folds.
Change in skin integrity | Baseline (T0), and change from baseline at twelve (T1), twenty (T2), and forty-eight (T3) weeks from baseline.
  effect of a light-to-moderate physical activity intervention on skin integrity, measured by videodermoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Giovanni Carta, MD, Principal Investigator — University of Cagliari
Locations (3):
- Italy (3):
  - Centro Obesità, AOU Cagliari, Cagliari
  - Clinica Dermatologica, AOU Cagliari, Cagliari
  - P.O. San Giovanni di Dio, AOU Cagliari, Cagliari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carta MG, Hardoy MC, Pilu A, Sorba M, Floris AL, Mannu FA, Baum A, Cappai A, Velluti C, Salvi M. Improving physical quality of life with group physical activity in the adjunctive treatment of major depressive disorder. Clin Pract Epidemiol Ment Health. 2008 Jan 26;4:1. doi: 10.1186/1745-0179-4-1. PMID 18221549
- [Result] Mura G, Carta MG. Physical activity in depressed elderly. A systematic review. Clin Pract Epidemiol Ment Health. 2013 Jul 12;9:125-35. doi: 10.2174/1745017901309010125. eCollection 2013. PMID 24009640
- [Result] Codella R, Luzi L, Inverardi L, Ricordi C. The anti-inflammatory effects of exercise in the syndromic thread of diabetes and autoimmunity. Eur Rev Med Pharmacol Sci. 2015 Oct;19(19):3709-22. PMID 26502862
- [Result] Rimland JM, Abraha I, Dell'Aquila G, Cruz-Jentoft A, Soiza R, Gudmusson A, Petrovic M, O'Mahony D, Todd C, Cherubini A. Effectiveness of Non-Pharmacological Interventions to Prevent Falls in Older People: A Systematic Overview. The SENATOR Project ONTOP Series. PLoS One. 2016 Aug 25;11(8):e0161579. doi: 10.1371/journal.pone.0161579. eCollection 2016. PMID 27559744
- [Result] Helmich I, Latini A, Sigwalt A, Carta MG, Machado S, Velasques B, Ribeiro P, Budde H. Neurobiological alterations induced by exercise and their impact on depressive disorders [corrected]. Clin Pract Epidemiol Ment Health. 2010 Nov 30;6:115-25. doi: 10.2174/1745017901006010115. PMID 21283646
- [Result] Mura G, Cossu G, Migliaccio GM, Atzori C, Nardi AE, Machado S, Carta MG. Quality of life, cortisol blood levels and exercise in older adults: results of a randomized controlled trial. Clin Pract Epidemiol Ment Health. 2014 Jun 13;10:67-72. doi: 10.2174/1745017901410010067. eCollection 2014. PMID 25006344
- [Result] Margraf J, Lavallee K, Zhang X, Schneider S. Social Rhythm and Mental Health: A Cross-Cultural Comparison. PLoS One. 2016 Mar 8;11(3):e0150312. doi: 10.1371/journal.pone.0150312. eCollection 2016. PMID 26954568
- [Result] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Pigliautile M, Ricci M, Mioshi E, Ercolani S, Mangialasche F, Monastero R, Croce MF, Federici S, Mecocci P. Validation study of the Italian Addenbrooke's Cognitive Examination Revised in a young-old and old-old population. Dement Geriatr Cogn Disord. 2011;32(5):301-7. doi: 10.1159/000334657. Epub 2012 Jan 19. PMID 22262124
- [Result] Monticone M, Baiardi P, Nava T, Rocca B, Foti C. The Italian version of the Sickness Impact Profile-Roland Scale for chronic pain: cross-cultural adaptation, reliability, validity and sensitivity to change. Disabil Rehabil. 2011;33(15-16):1299-305. doi: 10.3109/09638288.2010.527030. Epub 2010 Oct 29. PMID 21034202
- [Result] Dittmar M. Comparison of bipolar and tetrapolar impedance techniques for assessing fat mass. Am J Hum Biol. 2004 Sep-Oct;16(5):593-7. doi: 10.1002/ajhb.20066. PMID 15368607
- [Result] Paillard T, Pau M, Noe F, Gonzalez LM. Rehabilitation and Improvement of the Postural Function. Biomed Res Int. 2015;2015:703679. doi: 10.1155/2015/703679. Epub 2015 Nov 12. No abstract available. PMID 26640793
- [Result] Caronni A, Sterpi I, Antoniotti P, Aristidou E, Nicolaci F, Picardi M, Pintavalle G, Redaelli V, Achille G, Sciume L, Corbo M. Criterion validity of the instrumented Timed Up and Go test: A partial least square regression study. Gait Posture. 2018 Mar;61:287-293. doi: 10.1016/j.gaitpost.2018.01.015. Epub 2018 Jan 31. PMID 29413799
- [Result] Carruthers A, Carruthers J, Hardas B, Kaur M, Goertelmeyer R, Jones D, Rzany B, Cohen J, Kerscher M, Flynn TC, Maas C, Sattler G, Gebauer A, Pooth R, McClure K, Simone-Korbel U, Buchner L. A validated grading scale for forehead lines. Dermatol Surg. 2008 Nov;34 Suppl 2:S155-60. doi: 10.1111/j.1524-4725.2008.34364.x. PMID 19021673
- [Derived] Cossu G, Atzeni M, Cantone E, Forte V, Tusconi M, Kalcev G, Maleci A, Montisci R, Ferreli C, Atzori L, Primavera D, Dursun SM, Bert F, Tramontano E, Carta MG. Resilience to depression and unchanged quality of life in Sardinian old adults during COVID-19 lockdown. Front Psychiatry. 2025 Sep 3;16:1642413. doi: 10.3389/fpsyt.2025.1642413. eCollection 2025. PMID 40969700
- [Derived] Carta MG, Cossu G, Pintus E, Zaccheddu R, Callia O, Conti G, Pintus M, Aviles Gonzalez CI, Massidda MV, Mura G, Sardu C, Contu P, Minerba L, Demontis R, Pau M, Finco G, Cocco E, Penna MP, Orr G, Kalcev G, Cabras F, Lorrai S, Loviselli A, Velluzzi F, Monticone M, Cacace E, Musu M, Rongioletti F, Cauli A, Ruggiero V, Scano A, Crisafulli A, Cosentino S, Atzori L, Massa E, Mela Q, Fortin D, Migliaccio G, Machado S, Romano F, Preti A. Moderate Exercise Improves Cognitive Function in Healthy Elderly People: Results of a Randomized Controlled Trial. Clin Pract Epidemiol Ment Health. 2021 Sep 16;17:75-80. doi: 10.2174/1745017902117010075. eCollection 2021. PMID 34733346
- [Derived] Carta MG, Cossu G, Pintus E, Zoccheddu R, Callia O, Conti G, Pintus M, Gonzalez CIA, Massidda MV, Mura G, Sardu C, Contu P, Minerba L, Demontis R, Pau M, Finco G, Cocco E, Penna MP, Orru G, Kalcev G, Cabras F, Lorrai S, Loviselli A, Velluzzi F, Monticone M, Cacace E, Musu M, Rongioletti F, Cauli A, Ruggiero V, Scano A, Crisafulli A, Cosentino S, Atzori L, Massa E, Mela Q, Fortin D, Migliaccio G, Nardi AE, Angermeyer M, Preti A. Active elderly and health-can moderate exercise improve health and wellbeing in older adults? Protocol for a randomized controlled trial. Trials. 2021 May 7;22(1):331. doi: 10.1186/s13063-021-05278-6. PMID 33962664